CLINICAL TRIAL: NCT03264547
Title: A Phase III Clinical Study to Compare the Combination Therapy of Eribulin Mesylate + Pertuzumab + Trastuzumab With Paclitaxel or Docetaxel + Pertuzumab + Trastuzumab (EMERALD)
Brief Title: A Study to Compare Eribulin Mesylate + Pertuzumab + Trastuzumab With Paclitaxel or Docetaxel + Pertuzumab + Trastuzumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Breast Cancer Research Group (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRG-M06
Record Dates: First submitted 2017-08-01; First posted 2017-08-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Docetaxel; Paclitaxel; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Trastuzumab + pertuzumab + Taxane*
  *Taxane is chosen from the following; Docetaxel or Paclitaxel
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Docetaxel; Drug: Paclitaxel
- Arm B (Experimental): Trastuzumab+ Pertuzumab + Eribulin
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Eribulin

INTERVENTIONS:
Drug: Pertuzumab — Every 3 weeks
  Other Names: Perjeta
Drug: Trastuzumab — Every 3 weeks
  Other Names: Herceptin
Drug: Docetaxel — Every 3 weeks
  Other Names: Taxotere
  Arms: Arm A
Drug: Paclitaxel — Every week
  Other Names: Taxol
  Arms: Arm A
Drug: Eribulin — Administered for 2 weeks and is then stopped to be administered for 1 week
  Other Names: Halaven
  Arms: Arm B

SUMMARY:
To verify that combination therapy with trastuzumab + pertuzumab + eribulin brings similar PFS and better QOL compared to trastuzumab + pertuzumab + taxane in advanced/recurrent HER2-positive breast cancer patients who have no medical history of chemotherapy except ado-trastuzumab emtansine

ELIGIBILITY:
Inclusion Criteria:

1. Patients with breast cancer that is confirmed histologically or cytologically
2. Patients who are confirmed to be HER2 positive for the primary or a metastatic lesion at a participating medical institution
3. Patients with no medical history of treatment for advanced/recurrent cancer using a regimen of drugs including chemotherapeutics
4. >=6 months have passed since perioperative treatment with anticancer agents
5. Presence of a measurable lesion not required
6. Female aged 20-70 years old at the time of consent acquisition
7. Baseline left ventricular ejection fraction (LVEF) measured by ECHO or MUGA of >=50%
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
9. Patients who have maintained major organ functions, meeting all of the following criteria on a test within 28 days before enrollment. If there are multiple test results during this period, that obtained immediately before enrollment should be adopted.

(1) Neutrophil count: >=1,500/mm3 (2) Platelet count: >=100,000/mm 3 (3) Hemoglobin: >=9.0 g/dL (4) Total bilirubin: <=1.5 mg/dL (5) AST (GOT), ALT (GPT): <=2.5 times the ULN (<=5 times in those with liver metastasis) (6) Serum creatinine: <=1.5 mg/dL 10) Patients with a life expectancy of at least 6 months 11) Patient who submits written consent herself after receiving sufficient explanation about this study 12) Patients who can undergo QOL investigation

Exclusion Criteria:

1. Patients planning to undergo radical surgery if they respond to a treatment
2. Patients who have non-hematological adverse events assessed as Grade >=3 in the Common Terminology Criteria for Adverse Events ver. 4.0 in the Japanese JCOG version (CTCAE v4.0-JCOG) at the time of enrollment
3. Patients who have symptomatic metastases to the central nervous system or whose symptoms are hard to control
4. Patients who have active double cancer
5. Patients who have poorly controlled hypertension, or unstable angina
6. Patients who have a past history of congestive heart failure assessed as Class ll or higher in the New York Heart Association (NYHA) classification, or clinically significant arrhythmia requiring treatment
7. Patients with a past history of myocardial infarction within 6 months before enrollment
8. Patients who are expected to undergo major surgical treatment or who had severe injury within 28 days before enrollment, or who require major surgical treatment during the study treatment period
9. Patients with interstitial pneumonia which is symptomatic or requires treatment
10. Pregnant women, those with a positive pregnancy test, and lactating women
11. Patients with active systemic infection (including HCV and HBV), or who are found to be HIV-positive
12. Patients with hypersensitivity against pertuzumab and trastuzumab
13. Patients whom the investigator consider unable or unwilling to follow the protocol requirements

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
PFS | 5.75 years
  Progression-free survival

SECONDARY OUTCOMES:
RR | 5.75 years
  Response rate
DR | 5.75 years
  Duration of response
OS | 6.25 years
  Overall survival
PRO | 5.75 years
  Patient-reported outcomes(Numbness & tingling)
Safety | 5.75 years
  1. Incidence of infusion reactions and left ventricular dysfunction
  2. LVEF measurements during the study period
  3. Incidence and severity of adverse events and serious adverse events
  4. Abnormal laboratory test values
Biomaker | 5.75 years
  DNA mutation in the ctDNA and tumor tissue such as HER2,HER3, and PIK3CA
nMFS | 5.75 years
  new Metastases free survival
TTF of the subsequent treatment | 5.75 years
  Treatment duration of the following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Toshinari Tamashita, MD, PhD, Principal Investigator — Kanagawa Cancer Center; Norikazu Masuda, MD, PhD, Principal Investigator — NHO Osaka National Hospital; Shigehira Saji, MD, PhD, Principal Investigator — Fukushima Medical University
Locations (2):
- Japan (2):
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Background] Kaufman PA, Awada A, Twelves C, Yelle L, Perez EA, Velikova G, Olivo MS, He Y, Dutcus CE, Cortes J. Phase III open-label randomized study of eribulin mesylate versus capecitabine in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2015 Feb 20;33(6):594-601. doi: 10.1200/JCO.2013.52.4892. Epub 2015 Jan 20. PMID 25605862
- [Background] Wilks S, Puhalla S, O'Shaughnessy J, Schwartzberg L, Berrak E, Song J, Cox D, Vahdat L. Phase 2, multicenter, single-arm study of eribulin mesylate with trastuzumab as first-line therapy for locally recurrent or metastatic HER2-positive breast cancer. Clin Breast Cancer. 2014 Dec;14(6):405-12. doi: 10.1016/j.clbc.2014.04.004. Epub 2014 Jun 2. PMID 25024001
- [Derived] Yamashita T, Saji S, Takano T, Naito Y, Tsuneizumi M, Yoshimura A, Takahashi M, Tsurutani J, Iwatani T, Kitada M, Tada H, Mori N, Higuchi T, Iwasa T, Araki K, Koizumi K, Hasegawa H, Uchida Y, Morita S, Masuda N. Trastuzumab-Pertuzumab Plus Eribulin or Taxane as First-Line Chemotherapy for Human Epidermal Growth Factor 2-Positive Locally Advanced/Metastatic Breast Cancer: The Randomized Noninferiority Phase III EMERALD Trial. J Clin Oncol. 2025 Apr 10;43(11):1302-1313. doi: 10.1200/JCO-24-01888. Epub 2025 Jan 9. PMID 39787453
- [Derived] Yamashita T, Masuda N, Saji S, Araki K, Ito Y, Takano T, Takahashi M, Tsurutani J, Koizumi K, Kitada M, Kojima Y, Sagara Y, Tada H, Iwasa T, Kadoya T, Iwatani T, Hasegawa H, Morita S, Ohno S. Trastuzumab, pertuzumab, and eribulin mesylate versus trastuzumab, pertuzumab, and a taxane as a first-line or second-line treatment for HER2-positive, locally advanced or metastatic breast cancer: study protocol for a randomized controlled, non-inferiority, phase III trial in Japan (JBCRG-M06/EMERALD). Trials. 2020 May 7;21(1):391. doi: 10.1186/s13063-020-04341-y. PMID 32381018